CLINICAL TRIAL: NCT02036086
Title: A Pilot Study of the Neo-adjuvant Use of Vemurafenib Plus Cobimetinib (GDC-0973) in Patients With BRAF Mutant Melanoma With Palpable Lymph Node Metastases.
Brief Title: Study of Neo-adjuvant Use of Vemurafenib Plus Cobimetinib for BRAF Mutant Melanoma With Palpable Lymph Node Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28606
Record Dates: First submitted 2013-11-28; First posted 2014-01-14 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Melanoma stage IIIB or C with BRAF mutation; Recurrent regional lymphadenopathy not suitable for surgery; Eligible for neoadjuvant vemurafenib and cobimetinib
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vemurafenib, pill, twice daily (Experimental): Vemurafenib, 960 mg, oral, twice daily plus Cobimetinib, 60 mg, oral, four times daily
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib — Drug
  Other Names: Zelboraf
Drug: Cobimetinib — Drug
  Other Names: GDC-0973

SUMMARY:
This study will evaluate the clinical and pathological response to vemurafenib and cobimetinib in the neoadjuvant treatment of patients with histologically confirmed, BRAF V600 mutation-positive Stage IIIB and C melanoma. 20 patients will be treated with vemurafenib and cobimetinib for 2 months. Then they will be assessed for surgery. Patients will undergo surgery and subsequently resume taking vemurafenib and cobimetinib after recovery from surgery. Patients will undergo radiation therapy if appropriate then continue vemurafenib and cobimetinib. The maximum treatment period is 12 months. After 12 months of treatment, patients will be followed for disease recurrence and survival during for a total of 5 years.

DETAILED DESCRIPTION:
At Screening: Assessments will include CT or MRI of the brain, CT of chest, abdomen and pelvis, dermatology assessment, head and neck exam, pelvic and anal exam, ophthalmology exam, electrocardiogram (ECG), echocardiogram (ECHO) or multigated acquisition (MUGA) scan, a history and physical exam. A core biopsy will be performed within 14 days of study entry.

During Treatment: The maximum treatment period is 12 months. Patients will be assessed monthly while on treatment. Assessments performed will include vital signs assessment and physical exam, dermatology exam, ophthalmology exam, echocardiogram (ECHO) or multigated acquisition (MUGA) scan, electrocardiogram (ECG), safety blood tests, pelvic and anal exam.

Follow-up after treatment: Patients will be followed for 5 years. Radiology exams will be done to assess for disease. Other assessments performed include vital signs assessment and physical exam, dermatology exam, include echogram (ECHO) or multigated acquisition (MUGA) scans.

ELIGIBILITY:
Inclusion Criteria:

1. Naïve to treatment for locally advanced unresectable disease (Stage IIIB and C). Prior adjuvant therapy (including immunotherapy, e.g., ipilimumab) is allowed if prior to nodal recurrence and ≥ 3 months have elapsed from the last day of adjuvant therapy to start of study treatment.
2. Biopsy proven unresected melanoma patients with palpable regional lymph node metastases, presenting with AJCC stage IIIB-C or with recurrent regional lymphadenopathy that are not suitable or not preferred for surgical intervention.
3. BRAF V600 mutation positive.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
6. Adequate hematologic, renal and liver function within 7 days prior to the first dose of vemurafenib and cobimetinib.
7. Agree to always use an effective form(s) of contraception beginning from the informed consent signature date until at least 6 months after completion of study therapy.
8. Negative serum pregnancy test within 14 days prior to start of treatment in women of childbearing potential only.
9. Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

1. Cannot have received any prior therapy for the current recurrence or nodal disease. Previous adjuvant immunotherapy is allowed if prior to nodal recurrence and ≥ 3 months have elapsed from the last day of adjuvant therapy to start of study treatment.
2. History of prior RAF or MEK pathway inhibitor treatment.
3. Active malignancy (other than BRAF-mutated melanoma) or a previous malignancy within the past 3 years are excluded; except for patients with resected melanoma, resected basal cell carcinoma (BCC), resected cutaneous squamous cell carcinoma (SCC), resected melanoma in situ, resected carcinoma in-situ of the cervix, and resected carcinoma in-situ of the breast.
4. Evidence of distant metastatic disease.
5. History of clinically significant liver disease (including cirrhosis), current alcohol abuse, or known infection with Human Immunodeficiency Virus (HIV), hepatitis B virus, or hepatitis C virus.
6. Active infection or chronic infection requiring chronic suppressive antibiotics.
7. Pregnant or breastfeeding at the time of enrollment.
8. Active autoimmune disease (e.g., systemic lupus erythematosus, autoimmune vasculitis, inflammatory bowel disease [Crohn's disease and ulcerative colitis]).
9. Acromegaly
10. History of malabsorption or other clinically significant metabolic dysfunction.
11. Any other serious concomitant medical condition that would compromise safety or compromise the ability to participate in the study.
12. Requires a concomitant medication or dietary supplement that is prohibited during the study.
13. Unwillingness or inability to comply with study and follow-up procedures.
14. Current, recent (within 28 days of enrolment) or planned use of any investigational product outside of this study.
15. The following foods or supplements are prohibited at least 7 days prior to initiation of and during study treatment:

    1. St. John's wort or hyperforin
    2. Grapefruit juice
16. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment / central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration.
17. Currently are known to have the following conditions:

    1. Uncontrolled glaucoma with intra-ocular pressures with > 21 mmHg
    2. Retinal venous occlusion (RVO)
    3. Hypertensive retinopathy
18. Clinically significant cardiac dysfunction, including the following:

    1. Current unstable angina
    2. Current symptomatic congestive heart failure of New York Heart Association class 2 or higher
    3. History of congenital long QT syndrome or QTcF > 450 msec at baseline or uncorrectable abnormalities in serum electrolytes (sodium, potassium, calcium, magnesium, phosphorus).
    4. Current uncontrolled hypertension ≥Grade 2 (patients with a history of hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible).
    5. Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower.

17. Palliative radiotherapy or major surgery within 14 days prior to first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of treating patients with unresectable melanoma and palpable lymph node metastases that harbor the BRAF mutation with neoadjuvant vemurafenib. | 24 months

SECONDARY OUTCOMES:
Resectability rates post vemurafenib therapy | 5 years
Local-regional recurrence rates after treatment with neo-adjuvant vemurafenib. | 5 years
Time to distant metastases and Distant Metastatic Free Survival (DMFS). | 5 years
Disease Free Survival (DFS) and Overall Survival (OS). | 5 years
Immunohistochemical correlates of tumor response. | 5 years
Safety and tolerability of vemurafenib in the neoadjuvant setting | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Petrella, MD, BSc, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Balch CM, Soong SJ, Gershenwald JE, Thompson JF, Reintgen DS, Cascinelli N, Urist M, McMasters KM, Ross MI, Kirkwood JM, Atkins MB, Thompson JA, Coit DG, Byrd D, Desmond R, Zhang Y, Liu PY, Lyman GH, Morabito A. Prognostic factors analysis of 17,600 melanoma patients: validation of the American Joint Committee on Cancer melanoma staging system. J Clin Oncol. 2001 Aug 15;19(16):3622-34. doi: 10.1200/JCO.2001.19.16.3622. PMID 11504744
- [Background] Bevilacqua RG, Coit DG, Rogatko A, Younes RN, Brennan MF. Axillary dissection in melanoma. Prognostic variables in node-positive patients. Ann Surg. 1990 Aug;212(2):125-31. doi: 10.1097/00000658-199008000-00002. PMID 2375645
- [Background] Mocellin S, Pasquali S, Rossi CR, Nitti D. Interferon alpha adjuvant therapy in patients with high-risk melanoma: a systematic review and meta-analysis. J Natl Cancer Inst. 2010 Apr 7;102(7):493-501. doi: 10.1093/jnci/djq009. Epub 2010 Feb 23. PMID 20179267
- [Background] Hauschild A, Gogas H, Tarhini A, Middleton MR, Testori A, Dreno B, Kirkwood JM. Practical guidelines for the management of interferon-alpha-2b side effects in patients receiving adjuvant treatment for melanoma: expert opinion. Cancer. 2008 Mar 1;112(5):982-94. doi: 10.1002/cncr.23251. PMID 18236459
- [Background] Balch CM, Gershenwald JE, Soong SJ, Thompson JF, Atkins MB, Byrd DR, Buzaid AC, Cochran AJ, Coit DG, Ding S, Eggermont AM, Flaherty KT, Gimotty PA, Kirkwood JM, McMasters KM, Mihm MC Jr, Morton DL, Ross MI, Sober AJ, Sondak VK. Final version of 2009 AJCC melanoma staging and classification. J Clin Oncol. 2009 Dec 20;27(36):6199-206. doi: 10.1200/JCO.2009.23.4799. Epub 2009 Nov 16. PMID 19917835
- [Background] Shah GD, Socci ND, Gold JS, Wolchok JD, Carvajal RD, Panageas KS, Viale A, Brady MS, Coit DG, Chapman PB. Phase II trial of neoadjuvant temozolomide in resectable melanoma patients. Ann Oncol. 2010 Aug;21(8):1718-1722. doi: 10.1093/annonc/mdp593. Epub 2010 Jan 15. PMID 20080829
- [Background] Moschos SJ, Edington HD, Land SR, Rao UN, Jukic D, Shipe-Spotloe J, Kirkwood JM. Neoadjuvant treatment of regional stage IIIB melanoma with high-dose interferon alfa-2b induces objective tumor regression in association with modulation of tumor infiltrating host cellular immune responses. J Clin Oncol. 2006 Jul 1;24(19):3164-71. doi: 10.1200/JCO.2005.05.2498. PMID 16809739
- [Background] Gibbs P, Anderson C, Pearlman N, LaClaire S, Becker M, Gatlin K, O'Driscoll M, Stephens J, Gonzalez R. A phase II study of neoadjuvant biochemotherapy for stage III melanoma. Cancer. 2002 Jan 15;94(2):470-6. doi: 10.1002/cncr.10186. PMID 11900232
- [Background] Young K, Minchom A, Larkin J. BRIM-1, -2 and -3 trials: improved survival with vemurafenib in metastatic melanoma patients with a BRAF(V600E) mutation. Future Oncol. 2012 May;8(5):499-507. doi: 10.2217/fon.12.43. PMID 22646765
- [Background] Long GV, Menzies AM, Nagrial AM, Haydu LE, Hamilton AL, Mann GJ, Hughes TM, Thompson JF, Scolyer RA, Kefford RF. Prognostic and clinicopathologic associations of oncogenic BRAF in metastatic melanoma. J Clin Oncol. 2011 Apr 1;29(10):1239-46. doi: 10.1200/JCO.2010.32.4327. Epub 2011 Feb 22. PMID 21343559
- [Background] Sosman JA, Kim KB, Schuchter L, Gonzalez R, Pavlick AC, Weber JS, McArthur GA, Hutson TE, Moschos SJ, Flaherty KT, Hersey P, Kefford R, Lawrence D, Puzanov I, Lewis KD, Amaravadi RK, Chmielowski B, Lawrence HJ, Shyr Y, Ye F, Li J, Nolop KB, Lee RJ, Joe AK, Ribas A. Survival in BRAF V600-mutant advanced melanoma treated with vemurafenib. N Engl J Med. 2012 Feb 23;366(8):707-14. doi: 10.1056/NEJMoa1112302. PMID 22356324
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Background] Nazarian R, Shi H, Wang Q, Kong X, Koya RC, Lee H, Chen Z, Lee MK, Attar N, Sazegar H, Chodon T, Nelson SF, McArthur G, Sosman JA, Ribas A, Lo RS. Melanomas acquire resistance to B-RAF(V600E) inhibition by RTK or N-RAS upregulation. Nature. 2010 Dec 16;468(7326):973-7. doi: 10.1038/nature09626. Epub 2010 Nov 24. PMID 21107323
- [Background] Flaherty KT, Robert C, Hersey P, Nathan P, Garbe C, Milhem M, Demidov LV, Hassel JC, Rutkowski P, Mohr P, Dummer R, Trefzer U, Larkin JM, Utikal J, Dreno B, Nyakas M, Middleton MR, Becker JC, Casey M, Sherman LJ, Wu FS, Ouellet D, Martin AM, Patel K, Schadendorf D; METRIC Study Group. Improved survival with MEK inhibition in BRAF-mutated melanoma. N Engl J Med. 2012 Jul 12;367(2):107-14. doi: 10.1056/NEJMoa1203421. Epub 2012 Jun 4. PMID 22663011
- [Background] Larkin J, Ascierto PA, Dreno B, Atkinson V, Liszkay G, Maio M, Mandala M, Demidov L, Stroyakovskiy D, Thomas L, de la Cruz-Merino L, Dutriaux C, Garbe C, Sovak MA, Chang I, Choong N, Hack SP, McArthur GA, Ribas A. Combined vemurafenib and cobimetinib in BRAF-mutated melanoma. N Engl J Med. 2014 Nov 13;371(20):1867-76. doi: 10.1056/NEJMoa1408868. Epub 2014 Sep 29. PMID 25265494
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215